CLINICAL TRIAL: NCT01363063
Title: A Phase 1, Double-Blind, Study of the Tolerability of Formulations of Ketorolac Tromethamine Following Intranasal Administration in Healthy Volunteers
Brief Title: Study of the Tolerability of Ketorolac Tromethamine Following Intranasal Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ROX 2006-01
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ketorolac tromethamine (Part A) (Experimental)
  Interventions: Drug: Ketorolac tromethamine
- Ketorolac tromethamine (Part B) (Experimental)
  Interventions: Drug: Ketorolac tromethamine

INTERVENTIONS:
Drug: Ketorolac tromethamine — One dose of 15 mg ketorolac tromethamine with a lidocaine hydrochloride free formulation in one nostril and one dose of 15 mg ketorolac tromethamine containing 6% lidocaine hydrochloride in the other nostril
  Arms: Ketorolac tromethamine (Part A)
Drug: Ketorolac tromethamine — One dose of 15 mg ketorolac tromethamine containing 0% lidocaine hydrochloride into one nostril and either placebo or a single intranasal dose of 15 mg Ketorolac tromethamine containing 0%, 4% or 6% lidocaine hydrochloride into the other nostril
  Arms: Ketorolac tromethamine (Part B)

SUMMARY:
This was a Phase 1, double blind, two part study in healthy male and female volunteers. Each subject participated in only one part of the study. In Part A subjects received one dose of 15 mg ketorolac tromethamine with a lidocaine hydrochloride free formulation in one nostril and one dose of 15 mg ketorolac tromethamine containing 6% lidocaine hydrochloride in the other nostril, in a randomized manner. In Part B subjects were randomized to receive a single intranasal dose of 15 mg ketorolac tromethamine containing 0% lidocaine hydrochloride into one nostril and either placebo or a single intranasal dose of 15 mg ketorolac tromethamine containing 0%, 4% or 6% lidocaine hydrochloride into the other nostril. During the study, subjects remained resident from the morning of Day 1 until the afternoon of Day 1, when a post-study medical was performed prior to discharge.

The objective of this study was to compare the tolerability of formulations of ketorolac tromethamine with differing concentrations of lidocaine hydrochloride (0% and 6% in Part A and 0%, 4%, 6% and placebo in Part B) following intranasal administration to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, aged 18 to 60 years inclusive
* Female subjects of child bearing potential must have had a negative urine pregnancy test prior to entry into the study and must not have been breast feeding
* All female subjects of child bearing potential and all male subjects with female partners of child bearing potential must have consented to use a medically acceptable method of contraception (oral or implanted contraceptive hormones, condom or diaphragm with spermicidal agent, intrauterine device or surgical sterilization) throughout the study period
* Subject had given signed informed consent
* Subject was within 20% of normal weight for his/her height and body build according to the table of "Desirable Weights for Men and Women" (Metropolitan Life Insurance Co. 1999)
* Subject's medical history was considered normal, with no clinically significant abnormalities
* Subject was considered to be in good health in the opinion of the Investigator, as determined by a pre-study physical examination with no clinically significant abnormalities, vital signs within normal ranges and an electrocardiogram (ECG) with no clinically significant abnormalities
* Subject's pre-study clinical laboratory findings were within the normal range or if outside of the normal range were not deemed clinically significant in the opinion of the Investigator
* Subject had bilateral patent nasal airways at screening and Day 1 as assessed by the Investigator
* Body weight of at least 60 kg

Exclusion Criteria:

* Subject had had a clinically significant illness in the four weeks before screening
* Use of prescribed medications in the three weeks prior to dosing or over-the-counter preparations for seven days prior to dosing, except paracetamol which was allowed up to 48 hours prior to dosing. However, use of multivitamins and oral contraceptives were permitted
* Subject had a significant history of drug/solvent abuse, or a positive drugs of abuse test at screening
* Subject had a history of alcohol abuse or currently drank in excess of 28 units per week (males) or 21 units per week (females)
* Current tobacco use or a history of smoking within the past five years
* Subject was in the opinion of the Investigator not suitable to participate in the study
* Subject had participated in any clinical study with an investigational drug/device within three months prior to dosing
* Subject had a positive result of human immunodeficiency virus (HIV) screen, Hepatitis B screen or Hepatitis C screen
* Subject had had a serious adverse reaction or significant hypersensitivity to any drug
* Subject had donated 500 mL or more of blood within the three months prior to screening
* Any history of co-existing nasal polyps, NSAID sensitivity and asthma
* Allergic reaction to aspirin or other NSAIDs
* Current upper respiratory tract infection or other respiratory tract condition that could have interfered with the absorption of the nasal spray or with the assessment of adverse events (AEs)
* Any suspicion of rhinitis medicamentosa (chronic daily use of topical decongestants)
* Use of a monoamine oxidase inhibitor in the 14 days prior to study entry
* Active peptic ulcer disease, gastrointestinal bleeding or perforation, or a history of peptic ulcer disease or gastrointestinal bleeding
* Anemia due to unexplained or known gastrointestinal bleeding
* History of asthma or any other chronic pulmonary disorder
* Renal impairment or a risk of renal failure due to volume depletion
* Known sensitivity to lidocaine hydrochloride
* Previous history of nasal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12; Primary Completion 2007-02 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Discomfort Measurement on a Visual Analogue Scale | 15 minutes post-dose
  Following administration of each treatment, subjects completed a visual analogue scale (VAS) (ranging from "no discomfort" to "severe discomfort") at 1, 5, 10 and 15 minutes post-dose. If after the 15 minute VAS assessment discomfort was still present the subject was asked to complete further VAS assessments, at 5 minute intervals, until the discomfort had dissipated.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Clarke, BSc, MB BS, MFPM, Principal Investigator — ICON Developmental Solutions
Locations (1):
- ICON Developmental Solutions, Manchester, United Kingdom